CLINICAL TRIAL: NCT00417950
Title: Additional Glucose Lowering and Anti-Inflammatory Effects by Acarbose and Alcohol in Subjects With Impaired Glucose Tolerance or Mild Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Tri-Service General Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 950801/C06138
Record Dates: First submitted 2007-01-01; First posted 2007-01-04 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2007-01

CONDITIONS: Diabetes Mellitus; Impaired Glucose Tolerance
Keywords: diabetes; acarbose; alcohol; inflammation; oxidative stress; Mild diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Inflammation | interventions — Acarbose

INTERVENTIONS:
Drug: Acarbose

SUMMARY:
To understand if acarbose, an alpha-glucosidase inhibitor usually for treating diabetes, will further lower post meal glucose and inflammatory state when taking together with moderate amount of alcohol during meal tolerance test in subjects with impaired glucose tolerance or mild diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mild diabetes without prior medications or impaired glucose tolerance

Exclusion Criteria:

* Pregnancy
* Recent major cardiac, renal and hepatic disease
* Intolerance to alcohol
* Allergy to acarbose treatment

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2007-01

PRIMARY OUTCOMES:
Postprandial hyperglycemia

SECONDARY OUTCOMES:
Postprandial inflammatory responses
Postprandial oxidative stress

CONTACTS AND LOCATIONS:
Overall Officials: Wayne H Sheu, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan